CLINICAL TRIAL: NCT06980480
Title: A Multicenter, Randomized, Controlled, Open-label, Group-Sequential, Phase 3 Study to Investigate the Efficacy, Safety, and Tolerability of Intravenous Gammagard Liquid (Immune Globulin Infusion, 10%) for Primary Infection Prophylaxis Compared With Secondary Infection Prophylaxis in Adult Subjects With Multiple Myeloma Receiving B-Cell Maturation AntigenxCD3-Directed Bispecific Antibody Therapy
Brief Title: A Study of Gammagard Liquid (Immune Globulin Infusion, 10%) to Prevent Infections in Adults With Multiple Myeloma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry); Baxalta Innovations GmbH, now part of Takeda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TAK-339-3001; 2024-518420-80-00 (EU CTIS Number: EU CTIS Number)
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma; Secondary Immunodeficiency
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Primary Infection Prophylaxis: IGI, 10% (Experimental): Participants randomized to primary infection prophylaxis will receive a 400 milligrams per kilogram (mg/kg) dose of IGI, 10%, intravenously (IV) every 3 or 4 weeks within 3 days after randomization up to 12 months.
  Interventions: Biological: IGI, 10%
- Secondary Infection Prophylaxis: IGI, 10% (Active Comparator): Participants randomized to secondary infection prophylaxis will receive a 400 mg/kg dose of IGI, 10%, IV every 3 or 4 weeks only after experiencing at least one serious infection, as determined by the investigator, for the remainder of the 12 months observational period.
  Interventions: Biological: IGI, 10%

INTERVENTIONS:
Biological: IGI, 10% — IGI, 10% IV infusion.
  Other Names: TAK-339; Gammagard Liquid; KIOVIG

SUMMARY:
Multiple myeloma is a cancer of the plasma cells in the bone marrow.

The main aim of this study is to learn how well the Immune Globulin Infusion (human), 10 percentage (%) (IGI, 10%) can help prevent infections in participants with multiple myeloma receiving B-cell maturation antigen (BCMA) x cluster of differentiation 3 (CD3) directed bispecific antibody therapy.

Participants will be randomly assigned to one of two groups:

1. Primary infection prevention group: They will receive IGI, 10% for 12 months.
2. Secondary infection prevention group: They will only receive IGI, 10% if they develop a serious infection during the 12 months study period.

During the study, participants will visit their study clinic 15 times (for 4-week dosing interval) or 19 times (for 3-week dosing interval) and their total participation duration will be up to 14 months (including screening period of up to 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. The participants must have a documented diagnosis of Multiple Myeloma (MM) according to the guidelines by the International Myeloma Working Group (IMWG) before enrollment.
2. Participant who recently started teclistamab within the first 8 weeks of their planned treatment schedule and are planned to receive teclistamab for the next 12 months.
3. The participant or the participant's legally acceptable representative has provided informed consent (that is, in writing, documented via a signed and dated Informed Consent Form [ICF]) and any required privacy authorization before the initiation of any study procedures.
4. The participant is at least 18 years of age at the time of signing the ICF.
5. If a person of childbearing potential engages in sexual relations that carry risk of pregnancy, they agree to the following for the period from screening until 30 days after the last dose of study drug:

   1. To use a highly effective contraceptive method.
   2. To avoid donating ova.

Exclusion Criteria:

1. The participant has not achieved at least a minimal response to teclistamab within 8 weeks during the screening period.
2. The participant has a current serious infection or greater than (>) 1 serious infection in the past 3 months before screening.
3. The participant has a documented polyclonal IgG level less than (<) 150 milligrams per deciliter (mg/dL) at the most recent assessment before teclistamab initiation (within 4 weeks) as assessed by the investigator according to the site's standard practice.
4. The participant is currently receiving immunoglobulin products or has received immunoglobulin products within 16 weeks before screening.
5. The participant has received a hyperimmune or specialty high-titer immunoglobulin product (example, cytomegalovirus immune globulin, varicella-zoster immune globulin, hepatitis B immune globulin) within 30 days before screening.
6. The participant has received live viral vaccines within 30 days before screening.
7. The participant has an Eastern Cooperative Oncology Group performance status score of >2.
8. The participant has an active viral or bacterial infection or symptoms/signs of such an infection requiring treatment with anti-infectives within 1 week before enrollment.
9. The participant has received other B Cell Maturation Antigen (BCMA)*Cluster of Differentiation (CD3)-directed Bispecific Antibody therapy any time before screening.
10. The participant is scheduled to undergo plasmapheresis during the course of study or has undergone plasmapheresis in the last 16 weeks before screening.
11. The participant may be excluded from the study if, in the opinion of the investigator, the participant is at high risk for symptomatic hyperviscosity syndrome.
12. The participant has major surgery scheduled during the study, or the participant has not fully recovered from a recent major surgery (as judged by the investigator) during screening (participants with planned surgical procedures to be conducted under local anesthesia may participate).
13. The participant has an active secondary (non-MM) malignancy or other medical condition with life-expectancy of less than (<) 2 years.
14. The participant has a known history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) after Intravenous Immunoglobulin (IVIG) and/or immune serum globulin infusions.
15. The participant has a known history or current diagnosis of thromboembolic episodes such as deep vein thrombosis, pulmonary embolism, myocardial infarction, ischemic stroke, transient ischemic attack, peripheral artery disease within 6 months before screening.
16. The participant has moderate to severe renal dysfunction based on an estimated glomerular filtration rate less than or equal to (<=) 30 milliliters per minute per 1.73 square meters (mL/min/1.73 m^2), as defined by kidney disease: Improving Global Outcomes Clinical Practice Guideline for the Management of Glomerular Diseases, 2021 at the time of screening.
17. The participant has a known history of or is positive at screening for one or more of the following: hepatitis B surface antigen, Polymerase Chain Reaction (PCR) for hepatitis C virus, PCR for Human Immunodeficiency Virus (HIV) Type 1 and Type 2. Cured participants with a history of hepatitis C infection who have a negative PCR test at screening are eligible.
18. The participant has a documented diagnosis of a form of primary immunodeficiency (PID) involving a defect in antibody formation and requiring IgG replacement, as defined according to the International Union of Immunological Societies Committee.
19. The participant has a persistent serum aspartate aminotransferase and alanine aminotransferase >3.0 times the upper limit of normal at screening (may be repeated once to determine if it is persistent).
20. The participant has an immunoglobulin A (IgA) deficiency (<0.07 grams per liter [g/L]) with antibodies to IgA and a history of hypersensitivity reaction to IVIG.
21. Participant with a known systemic hypersensitivity to any of the excipients of IGI, 10% in accordance with the investigator's brochure/package insert/Summary of Product Characteristics.
22. Known substance abuse including opiates, psychostimulant agents, or other illicit drugs with the exception of cannabinoids within 12 months of screening.
23. The participant has anemia that would preclude phlebotomy for laboratory studies, according to standard practice at the site, at the discretion of the investigator (may be repeated once to determine if it has resolved).
24. The participant has a medical condition, laboratory finding, or physical examination finding that precludes participation or with clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may interfere with the successful completion of the study or place the participant at undue medical risk.
25. The participant is receiving immunosuppressive treatment (other than for MM or corticosteroids) at screening or plans to receive immunosuppressive treatment after study enrollment.
26. The participant or the participant's legally designated representative is not willing and able to comply with the protocol requirements.
27. The participant has participated or is scheduled to participate in another clinical study involving an investigational product (IP) or investigational device within 30 days before screening and during the course of the study.
28. The participant is a family member or employee of the investigator or the investigator's site staff.
29. The participant is pregnant or has a positive pregnancy test or is lactating at the time of screening or enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2028-09-11 (Estimated); Study Completion 2028-09-11 (Estimated)

PRIMARY OUTCOMES:
Time To the First Serious Infection | Up to 12 months

SECONDARY OUTCOMES:
Number of Participants With at Least 1 Serious Infection | Up to 12 months
Annualized Rate of Days on Antibiotics for Treatment of Bacterial Infections | Up to 12 months
Annualized Rate of Bacterial Infections | Up to 12 months
Annualized Rate of Serious Infections | Up to 12 months
Annualized Rate of Acute Serious Bacterial Infections (ASBIs) | Up to 12 months
Number of Participants With Any Infections | Up to 12 months
Duration of Infections | Up to 12 months
Time To Any First Infection | Up to 12 months
Annualized Rate of Any Infections | Up to 12 months
Number of Participants With Bacterial/Viral Infection/Fungal Infection | Up to 12 months
  Number of participants with bacterial/viral infection, including covid/fungal infection diagnosed clinically and via microbiology (culture, polymerase chain reaction [PCR], other imaging will be reported.
Annualized Rate of Episodes of Fever due to Infections | Up to 12 months
Total Immunoglobulin G (IgG) Levels in Serum | 3-Week dosing: Day 1 up to Day 357; 4-Week dosing: Day 1 up to Day 364
IgG Subclasses (IgG1, IgG2, IgG3, and IgG4) Levels in Serum | 3-Week dosing: Day 1 up to Day 357; 4-Week dosing: Day 1 up to Day 364
Antigen-specific Antibody Levels in Serum | 3-Week dosing: Day 1 up to Day 357; 4-Week dosing: Day 1 up to Day 364
Number of Participants With Adverse Event (AEs) and Treatment-Emergent Adverse Events (TEAEs) | Up to 12 months
Number of Participants With TEAEs Related to IGI, 10% | Up to 12 months
Number of Participants With TEAEs Temporally Associated to the IGI, 10% Within 72 hours of Administration | Within 72 hours of IGI, 10% administration (up to 12 months)
Number of Participants With Infusion Withdrawals, Interruptions, and Infusion Rate Reductions due to TEAEs Related to IGI, 10% | Up to 12 months
Number of Participants With at Least 1 Hospitalization due to Infection | Up to 12 months
Number of Hospitalizations, Including Intensive Care Unit (ICU) and Non-ICU due to Infection | Up to 12 months
Number of Participants With Outpatient Visits, Including Emergency Room (ER) Visits due to Infection | Up to 12 months
Duration of Hospitalizations, Including ICU and Non-ICU due to Infection | Up to 12 months
Number of Days of Hospitalization per Participant-year, Including ICU and Non-ICU due to Infection or Other Reasons | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (16):
- United States (9):
  - Infirmary Health - Diagnostic & Medical Clinic (DMC), Mobile, Alabama
  - Chao Family Comprehensive Cancer Center UCI, Orange, California
  - University of Kansas, Westwood, Kansas
  - University of Maryland | Greenebaum Cancer Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New York Oncology Hematology, Albany, New York
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
- United Kingdom (7):
  - Royal Devon And Exeter Hospital, Exeter, Devon
  - Colchester General Hospital, Colchester, Essex
  - Gloucestershire Royal Hospital, Gloucester, Gloucestershire
  - Cardiff & Vale University Health Board, Cardiff, South Glamorgan
  - Harrogate and District NHS Foundation Trust, Harrogate
  - Milton Keynes University Hospital NHS Foundation Trust, Milton Keynes
  - County Hospital (Stafford Hospital), Stafford

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/0507a411bcd348ca??page=1&idFilter=TAK-339-3001